CLINICAL TRIAL: NCT05052125
Title: Substudy: Oxygen Therapy in COPD Patients - Oxidative Stress and Mortality
Brief Title: Substudy of Protocol 2019-002498-80 - NCT04223050: Comparing Mortality for Low vs High Peripheral Oxygen Saturation in COPD-patients With Acute Exacerbation (O2flow-COPD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of inclusion of patients
Sponsor: Mikkel Brabrand (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Mikkel Brabrand, Professor, ph.d., MD, Esbjerg Hospital - University Hospital of Southern Denmark
Organization: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002498-80 substudy
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: oxygen; oxidative stress; mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High oxygen saturation (Active Comparator): Peripheral oxygen saturation level >94% Intervention: Drug: Oxygen gas
  Interventions: Drug: Oxygen
- Low oxygen saturation (Active Comparator): Peripheral oxygen saturation level 88-92% Intervention: Drug: Oxygen gas
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Administering oxygen to achieve the desired peripheral oxygen saturation

SUMMARY:
As protocol NCT04223050. This substudy furthermore investigates the role of oxidative stress in the administration of oxygen in COPD patients.

DETAILED DESCRIPTION:
Studies have shown that oxidative stress plays a critical role in the pathogenesis of COPD and its comorbidities. Oxidative stress refers to a state in which the activity of oxidants (e.g. reactive oxygen species (ROS)) outweighs that of antioxidants. ROS can be introduced exogenously by for example cigarette smoke and atmospheric pollution, but is also produced endogenously as a byproduct of ATP production in mitochondria or from immune cells during oxidative burst. When high fractions of inspired oxygen are administered, excess O2 can lead to formation of additional ROS, which depletes antioxidants and induces an inflammation with leukocyte-derived inflammatory mediators migrating to the site of injury. In turn, this causes cellular hypertrophy, increased surfactant secretion, and cellular influx of monocytes and mast cells. During the final, fibrotic phase of oxygen toxicity, irreversible, persistent destruction of the pulmonary lining have occurred with collagen disposition, thickening of pulmonary interstitial space, and fibrosis.

This substudy therefore aim to investigate the relation between oxygen therapy in COPD patients admitted with acute exacerbation, oxidative stress, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* ability to give informed consent
* previously diagnosed COPD (either confirmed diagnosis at prior hospital - contact or from their general practitioner or confirmed diagnosis by the treating physician in the emergency department (verified by use of relevant medication))
* admitted with acute exacerbation (acute and worsened shortness of breath) of COPD
* requiring oxygen treatment

Exclusion Criteria:

* Instability at arrival requiring immediate lifesaving treatment, e.g. intubation or non-invasive ventilation, within the first 30 minutes
* Expected total length of stay in hospital < 12 hours
* Planned transfer to another hospital within 12 hours
* Unwilling to have repeated arterial blood gas analyses within the first 12 hours
* Patients judged terminal by treating physician in the emergency department
* Non-residents of the particular country
* Expected impossible follow-up
* Fertile women (<50 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Prior participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Oxidative stress levels (systemic and lung 8-isopropane levels). | Immediately after study completion

SECONDARY OUTCOMES:
Inflammation levels (systemic and lung IL-8 levels) | Immediately after study completion
7-day all-cause mortality and 30-day all-cause mortality | 30 days
  extracted from the Danish national registries
over-all length of hospital stay | Immediately after study completion
  calculated from the hospital records
respiratory acidosis | Immediately after the procedure
  measured as an arterial blood gas analysis with pH < 7.35 and hypercapnia

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hospital of Southern Denmark, Esbjerg, Esbjerg
  - Kolding Hospital, Sygehus Lillebælt, Kolding

IPD SHARING:
Plan to Share IPD: No